CLINICAL TRIAL: NCT02053675
Title: Hemodynamic Effects of Low Doses of Arginine Vasopressin in Early Septic Shock Stage
Brief Title: Hemodynamic Effects of Vasopressin in Early Septic Shock Stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Vasopress FAPESP 2010/50096-6
Record Dates: First submitted 2013-05-28; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2010-05

CONDITIONS: Septic Shock
Keywords: septic shock; vasopressin; microcirculation; tissue oxygenation; vasopressors; hemodynamics
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vasopressin (Other)
  Interventions: Drug: Vasopressin infusion

INTERVENTIONS:
Drug: Vasopressin infusion

SUMMARY:
Vasopressin is a vasopressor used in patients with septic shock. However, its systemic hemodynamic effects and its microcirculation effects are not completely known and understood. This study aimed to evaluate the effect of exogenous vasopressin on sublingual microcirculation using the sidestream dark field technique and to correlate it with its systemic effects. To this prospective interventional study, patients with septic shock were included during the first 48 hours of use of catecholamine vasopressors, admitted to the intensive care unit of a university hospital. Vasopressin was administered at 0.04 U / min for one hour. Systemic hemodynamic measurements were obtained immediately before and 1 hour after vasopressin. In addition, images of sublingual microcirculation were collected through sidestream dark field technology. Further analysis with specific software was done after.

DETAILED DESCRIPTION:
Immediately before vasopressin infusion, fluid responsiveness was evaluated by delta PP (ΔPP) with ΔPP module attached to the monitor (DX 20x20, Dixtal, São Paulo, Brazil). Continuous sedation was maintained to control spontaneous ventilatory efforts. ΔPP > 13% receive crystalloid (Ringer's lactate or normal saline 0.9%) challenges until the ΔPP were below this value. Patients in whom was not possible to measure ΔPP, received crystalloid aliquots of 500 ml until there was no increase in cardiac output greater than 10%. Vasopressors were used to maintain mean arterial pressure above 65 mmHg. The fraction of inspired oxygen was adjusted to maintain oxygen saturation between 92-94%.

Thirty minutes after initial stabilization (the pre-vasopressin), all hemodynamic and respiratory measurements were obtained (pre-vasopressin), namely mean arterial pressure (MAP), heart rate (HR), right atrial pressure (RAP) , mean pulmonary artery pressure (MPAP), occluded pulmonary artery pressure (OPAP), cardiac index (CI), stroke index (SI), systemic vascular resistance index (SVRI), pulmonary vascular resistance index (PVRI). Samples were collected for blood gas analysis and arterial and mixed venous blood lactate.

Direct analysis of the sublingual microcirculation was done at that time by videomicroscopy obtained by SDF (Microscan; MicroVision Medical, Amsterdam, Netherlands), following the protocol previously described. Briefly, after removal of secretions, the lens of SDF was placed in the sublingual space without exerting any pressure. All images were obtained by a qualified physician using the recommended techniques to ensure image quality. We obtained three sequential images of high quality stable for at least 20 seconds, of both sides of the tongue while avoiding artifacts pressure. All images were captured using a notebook and a video converter analog / digital (ADVC110, Canopus Co, San Jose, California).

After obtaining baseline data, vasopressin was infused at fixed dose of 0.04 U / min. After one hour of vasopressin(post-vasopressin), the same variables were collected. If required, the adrenergic vasopressors infusion was adjusted during the study to maintain the target MAP from 65 to 70 mmHg. If patients were receiving dobutamine, its dose was kept constant during the study procedures. If fluid replacement or adjustment of ventilatory parameters or sedation were needed during the study, the patient was excluded.

All images were subsequently analyzed using the AVA 3.0 ® software (Microvision Medical, Amsterdam, Netherlands), considering only vessels with a diameter less than 20 micrometers. A blinded investigator analyzed all the images in a random order. The microcirculatory flow index (MFI), the total vascular density (TVD), the proportion of perfused vessels (PPV), the perfused vessel density (PVD), and the heterogeneity index (HI) were calculated.

Briefly, the MFI is calculated from the imaginary division of the image captured and stabilized into four quadrants. Its calculation is the average of the subjective evaluation of the flow in the four quadrants, quantified 0-3, where 0 corresponds to absent flow, 1 intermittent flow, 2 and 3 sluggish flow and continuous flow, respectively. TVD is calculated from the assumption that it is proportional to the number of vessels crossing three horizontal lines and three vertical equidistant arbitrary placed in the overlay image. The program computes the number of vessels crossing the lines and vessels and the total is divided by the lines length. Perfusion subjective evaluation was done in each vessel, graduated from 0 to 3 (absent, intermittent, sluggish or continuous). The PPV is calculated from the total number of vessels counted in the TVD subtracted not perfused vessels (those with flow 0 or flow 1), according to the formula: PPV = TVD - not perfused vessels / TVD x100. The PVD is obtained by multiplying TVD and PPV. The HI is calculated from the difference between the highest and lowest MFI found in three images captured in each moment (before and after vasopressin), according to the formula: HI = highest MFI - lowest MFI / MFI average.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Septic shock using adrenergic vasopressors for less than 48 hours
* Arterial catheter and pulmonary artery catheter with semi measurement of cardiac output by thermodilution (Vigilance, Edwards Lifesciences, Irvine, CA, USA) inserted
* Signed consent declaration

Exclusion Criteria:

* Acute coronary disease
* Suspected or confirmed acute mesenteric ischemia
* Severe hyponatremia (Na + <130 mmol / L)
* Raynaud's phenomenon
* Sclerodermia
* Pregnancy
* Technical difficulties to capture videomicroscopy with sublingual SDF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to evaluate the effect of vasopressin infusion in microcirculation of septic shock patients | one hour after vasopressin initiation
  Significant changes in microcirculatory parameters - MFI (absolute number), TVD (mm/mm2), PVD (mm/mm2), PPV (%), HI (%)

SECONDARY OUTCOMES:
The secondary objectives were to evaluate the effects of vasopressin on macrocirculation, and correlate potential microcirculatory effects related to its use, with baseline systemic circulation and microcirculation. | one hour after vasopressin initiation
  Significant changes in HR (bpm), CI (L/min.m2), SI (ml/beat/m2), oxigen delivery (ml/min), lactate (mg/dL), CO2 gradient (mmHg), and correlation between these changes and potential microcirculatory parameters alteration (MFI, TVD, PVD, PPV, HI)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital São Paulo, São Paulo, São Paulo/SP, Brazil

REFERENCES:
- [Derived] Nascente APM, Freitas FGR, Bakker J, Bafi AT, Ladeira RT, Azevedo LCP, Lima A, Machado FR. Microcirculation improvement after short-term infusion of vasopressin in septic shock is dependent on noradrenaline. Clinics (Sao Paulo). 2017 Dec;72(12):750-757. doi: 10.6061/clinics/2017(12)06. PMID 29319721